CLINICAL TRIAL: NCT00326183
Title: An Open, Multicenter Study of the Safety and Tolerability of VAQTA(TM) and ProQuad(TM) in Healthy Children 12 to 23 Months of Age
Brief Title: Hepatitis A Vaccine, Inactivated and Measles, Mumps, Rubella and Varicella Virus Vaccine Live Safety Study (V251-066)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V251-066; 2006_023
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Results first posted 2008-11-20 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis A; Measles; Mumps; Rubella; Chickenpox
MeSH Terms: conditions — Hepatitis A; Measles; Mumps; Rubella; Chickenpox | interventions — Hepatitis A Vaccines; measles, mumps, rubella, varicella vaccine

ARMS (2):
- 1 (Active Comparator): Arm 1: vaccine
  Interventions: Biological: VAQTA®
- 2 (Active Comparator): Arm 2: Active comparator
  Interventions: Biological: VAQTA®; Biological: ProQuad

INTERVENTIONS:
Biological: VAQTA® — 0.5 ml injection VAQTA®; 2nd 0.5 ml injection VAQTA® 24 week period of treatment.
  Other Names: V251
Biological: ProQuad — 0.5 ml injection ProQuad; 2nd 0.5 ml injection ProQuad®. 24 week period of treatment.
  Arms: 2

SUMMARY:
Two doses each of Hepatitis A Vaccine, Inactivated and Measles, Mumps, Rubella and Varicella [Oka/Merck] Virus Vaccine Live will be given concomitantly or non-concomitantly. Safety data will be collected following each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Negative clinical history of hepatitis A, measles, mumps, rubella, varicella (chickenpox), and/or zoster
* No other vaccinations scheduled to be administered at the time of the first or second doses of VAQTA(TM) and ProQuad(TM)

Exclusion Criteria:

* Previously vaccinated with any hepatitis A vaccine, measles, mumps, rubella, and/or varicella vaccine either alone or in any combination
* History of allergy to any vaccine component
* History of seizure disorder
* Immunosuppressed including congenial and acquired conditions and immunosuppressive therapy
* Known severe thrombocytopenia or any other coagulation disorder that would contraindicate intramuscular injections
* Recent (<72 hours) febrile illness (>100.3 degrees F [>37.9 degrees C] oral equivalent) prior to study vaccination.

Ages: 12 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Actual)
Dates: Start 2007-03-26 (Actual); Primary Completion 2008-01-15 (Actual); Study Completion 2008-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Petrecz M, Acosta CJ, Klopfer SO, Kuter BJ, Goveia MG, Stek JE, Schodel FP, Lee AW. Safety and immunogenicity of VAQTA(R) in children 12-to-23 months of age with and without administration of other US pediatric vaccines. Hum Vaccin Immunother. 2019;15(2):426-432. doi: 10.1080/21645515.2018.1530934. Epub 2018 Nov 15. PMID 30431383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 investigators in the United States; Date of first subject visit: 26-Mar-2007.
  Date of last subject visit: 14-Nov-2007.
Groups:
- Arm 1: VAQTA™: Hepatitis A vaccine, inactivated
- Arm 2: VAQTA™ +ProQuad™: Hepatitis A vaccine, inactivated + measles, mumps, rubella, and varicella vaccine live
Period: Overall Study
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Started | 1453 | 347
Vaccination 1 + Safety Follow-up | 1453 | 347
Postvaccination 1 Post-safety Follow-up | 1393 | 325
Vaccination 2 + Safety Follow-up | 1301 | 292
Postvaccination 2 Post-safety Follow-up | 1265 | 271
Completed | 1253 | 264
Not Completed | 200 | 83
Not completed — Lost to Follow-up | 104 | 56
Not completed — Protocol Violation | 6 | 3
Not completed — Withdrawal by Subject | 35 | 7
Not completed — Subject Moved | 7 | 4
Not completed — Other | 47 | 13
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™ | Total
Number analyzed (Participants) | 1453 | 347 | 1800
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.3 (1.49) | 12.5 (0.90) | 13.2 (1.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 703 | 176 | 879
  Male | 750 | 171 | 921

OUTCOME MEASURES:

1. Primary Outcome: Participants With 1 or More Serious Vaccine-Related Adverse Experiences
Time Frame: Days 1 to 14 after any vaccination
Population: Includes all subjects who provided safety follow-up data after any dose of vaccine out of the total number of subjects enrolled.
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 1415 | 334
participants | 0 | 1

2. Secondary Outcome: Participants With 1 or More Systemic Adverse Experiences
Time Frame: Days 1 to 14 After Any Vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 1415 | 334
participants | 782 | 197

3. Primary Outcome: Participants With 1 or More Injection-Site Adverse Experiences
Time Frame: Days 1 to 14 after any vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 1415 | 334
participants | 701 | 164

4. Primary Outcome: Participants With Measles-Like Rash After First Vaccination
Time Frame: Days 1 to 28 After First Vaccination
Population: Includes all subjects who provided safety follow-up data after the first vaccinations were administered. Only the VAQTA™ +ProQuad™ group was followed for rashes.
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 0 | 328
participants |  | 13

5. Primary Outcome: Participants With Measles-Like Rash After Second Vaccination
Time Frame: Days 1 to 28 After Second Vaccination
Population: Includes all subjects who provided safety follow-up data after the second vaccinations were administered. Only the VAQTA™ + ProQuad™ group was followed for rashes.
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 0 | 263
participants |  | 5

6. Primary Outcome: Participants With Mumps-Like Symptoms After First Vaccination
Time Frame: Days 1 to 28 After First Vaccination
Population: Includes all subjects who provided safety follow-up data after the first vaccinations were administered. Only the VAQTA™ + ProQuad™ group was followed for mumps-like symptoms.
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 0 | 328
participants |  | 0

7. Primary Outcome: Participants With Mumps-Like Symptoms After Second Vaccination
Time Frame: Days 1 to 28 After Second Vaccination
Population: Includes all subjects who provided safety follow-up data after the second vaccinations were administered. Only the VAQTA™ + ProQuad™ group was followed for mumps-like symptoms.
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 0 | 263
participants |  | 0

8. Primary Outcome: Participants With Rubella-Like Rash After First Vaccination
Time Frame: Days 1 to 28 After First Vaccination
Population: Includes all subjects who provided safety follow-up data after the first vaccinations were administered. Only the VAQTA™ + ProQuad™ group was followed for rashes.
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 0 | 328
participants |  | 1

9. Primary Outcome: Participants With Rubella-Like Rash After Second Vaccination
Time Frame: Days 1 to 28 After Second Vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 0 | 263
participants |  | 0

10. Primary Outcome: Participants With Varicella/Zoster-Like Rash After First Vaccination
Time Frame: Days 1 to 28 After First Vaccination
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 0 | 328
participants |  | 0

11. Primary Outcome: Participants With Varicella/Zoster-Like Rash After Second Vaccination
Time Frame: Days 1 to 28 After Second Vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 0 | 263
participants |  | 0

12. Primary Outcome: Participants With Elevated Temperature (>=102.2F/39.0C)
Time Frame: Days 1 to 5 After Any Vaccination
Population: Includes all subjects who provided body temperature follow-up data after any dose of vaccine.
Measure: Number; unit: participants
Arm/Group | Arm 1: VAQTA™ | Arm 2: VAQTA™ +ProQuad™
Number analyzed (Participants) | 1383 | 320
participants | 56 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.